CLINICAL TRIAL: NCT03362840
Title: Integrating the Early Started Denver Model in Israeli Autism Spectrum Disorder Preschools: A Controlled Trial
Brief Title: Integrating the ESDM in ASD Preschools in Israel
Acronym: ESDM-ISR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bar-Ilan University, Israel (Other)
Collaborators: Association for Children at Risk (Other)
Responsible Party: Principal Investigator, Ofer Golan, Prof., PhD, Bar-Ilan University, Israel
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: BarIlanU
Record Dates: First submitted 2017-11-30; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Start Denver Model (ESDM) group (Experimental): The ESDM is a manualized comprehensive treatment model for young children (12-48 months). In the preschool based ESDM, learning objectives are guided by the ESDM curriculum checklist, which includes developmental skills in language, play, motor skills, personal independence, imitation and cognition.
  Interventions: Behavioral: Early Start Denver Model
- Eclectic preschool intervention group (Active Comparator): The eclectic approach consists of a combination of methods from several treatment-models. Individualized educational plans are based on multi-disciplinary assessment, and include objectives in several domains - communication, social-skills, play, emotional adjustment, adaptive daily skills, motor skills and cognition. They are presented to parents at the beginning of the year and are reviewed by the staff three times a year.
  Interventions: Behavioral: Eclectic preschool intervention

INTERVENTIONS:
Behavioral: Early Start Denver Model — The ESDM is a manualized comprehensive treatment model for young children (12-48 months). In the preschool based ESDM, learning objectives are guided by the ESDM curriculum checklist, which includes developmental skills in language, play, motor skills, personal independence, imitation and cognition. The objectives are monitored for progress during each session The sessions are conducted according to ESDM principles, and include weekly parent-coaching session, in which parents observe the therapist interact with the child while applying various teaching techniques, and then implement these techniques during the interaction with their child. Additionally, parents get acquainted with the daily objective sheet and are encouraged to work on these objectives at home as well. Finally, in this model, therapist adherence to the ESDM practices are monitored according to the ESDM fidelity rating system
  Arms: Early Start Denver Model (ESDM) group
Behavioral: Eclectic preschool intervention — The eclectic approach consists of a combination of methods from several treatment-models. Individualized educational plans are based on multi-disciplinary assessment, and include objectives in several domains - communication, social-skills, play, emotional adjustment, adaptive daily skills, motor skills and cognition. They are presented to parents at the beginning of the year and are reviewed by the staff three times a year.
  Parents attend by-weekly counseling-sessions with a professional in order to receive input regarding their child's progress, and discuss issues concerning their child's functioning. All staff members receive supervision at various intensities. However, these usually do not adhere to a single structure and are not guided by official fidelity criteria.
  Arms: Eclectic preschool intervention group

SUMMARY:
The current study evaluates the effectiveness of the Early Start Denver Model (ESDM) when integrated in existing community preschools for children with ASD. The study compares developmental gains made a group of children receiving preschool-based ESDM compared to a group of children receiving eclectic interventions in their preschools (treatment as usual).

DETAILED DESCRIPTION:
The Early Start Denver Model is a comprehensive treatment model for young children with Autism Spectrum Disorders (ASD), which builds upon behavioral, relationship, play-based and developmental theories and practices. Utilizing the plasticity of the young brain, while managing social attention, employing multi-modal teaching, and tapping into the child's motivation, the ESDM aims to alter the child's developmental trajectories by creating rich and meaningful learning experiences in daily and naturalistic routines. This model focuses on all areas of development, with significant stress on communication, language, social skills, play and imitation. In the ESDM, parents are seen as a main motivational factor for the child, and a focal part in planning and implementing key components of the intervention.

Currently, community preschool settings are the main providers of intervention programs for children with ASD in Israel. The prevalent mode of intervention in these settings is a multi-disciplinary eclectic model, in which professionals from various disciplines deliver intervention comprising several theories and practices. While quite ubiquitous, this type of intervention was shown in previous research as less effective than specialized, comprehensive treatment models.

The ESDM was previously shown efficacious in intensive home-based delivery, and effective as a center-based group model. However, there are currently no studies that assess the effectiveness of the ESDM when integrated in existing community preschool settings. Additionally, previous research in center-based group delivery of the ESDM did not focus on the effects of routine parental involvement in child treatment (when delivered in a preschool setting) on child and parental outcomes. The current study aims to explore the effects of ESDM implementation in community preschool settings, together with incorporation of parents in the treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Children learning in ASD schools with a diagnosis of ASD validated by the Autism Diagnostic Observation Schedule - 2nd edition.
* ESDM group: parents who have agreed to participate in weekly joint sessions at the preschool.

Exclusion Criteria:

-

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Mullen Scales of Early Learning (MSEL) | Pre-intervention, 8 months, 20 months
  A standardized measure of early development which is administered to children from birth to 68 months of age. The MSEL includes five subscales: receptive language, expressive language, visual reception, fine motor, and gross motor skills, for which a standard T score and age equivalents (AE) are computed, together with a total composite of intellectual ability. Administration time - 30-60 minutes (Mullen, 1995).
Change from baseline Vineland Adaptive Behavior Scales, Second Edition (VABS-II) | Pre-intervention, 8 months, 20 months
  A structured interview measuring adaptive behavior from birth to adulthood. This measure is divided into 11 sub-scales, clustered into four domains: communication, daily living skills, socialization and motors skills. Standard scores and age equivalents can be obtained from this measure, together with an adaptive behavior composite (ABC). The VABS-II may be administered via a structured interview with the caregiver or teacher, or using a self-report questionnaire filled out by the responder. In the current study, both forms of administration will be used, so that parents will be interviewed by a trained practitioner, and teachers will be given the self-report version of the test. Administration time - 45-60 minutes (Sparrow, Cicchetti & Balla, 2005).

SECONDARY OUTCOMES:
Change from baseline Parent Sense of Competence Scale (PSOC) | Pre-intervention, 8 months, 20 months
  A 16 item self- report questionnaire designed to measure parental sense of efficacy and satisfaction in parenting. The 16 items of the inventory are rated on a 6 point Likert scale, with higher scores indicating to higher sense of efficacy and satisfaction. The PSOC was reported by the authors to have adequate internal reliability for both subscales. Additionally, the PSOC was found to be negatively correlated with measures of child behavior problems (Johnston & Mash, 1989).
Change from baseline Parenting Stress Index - Short Form (PSI\SF) | Pre-intervention, 8 months, 20 months
  A 36 item questionnaire assessing parenting distress, parent-child dysfunctional interactions, and perception of child as difficult to manage. Items are rated on a 5 point Likert scale, with higher scores pointing to higher parental stress. The PSI\SF (Abidin, 1995) was used in several studies assessing stress in parents to children with autism, and was reported to have high internal consistency and test-retest reliability (for example, Davis-Ornstein & Carter, 2008; Hall & Graff, 2011).
Change from baseline parent-child interaction paradigm | Pre-intervention, 8 months, 20 months
  In this paradigm, parents and children will be video-recorded during a 7 minute free-play interaction, in order to assess changes in child social-communication, play and restrictive-repetitive behaviors, and parental interactive behaviors. The video-records will be then coded micro-analytically using the Noldus Observer software, to capture moment to moment changes in child-parent interaction measures.
Change from baseline child-staff member interaction paradigm | Pre-intervention, 8 months, 20 months
  In this paradigm, the child will be video recorded with a staff member from his preschool during 7 minutes of free play, in order to measure child social-communication, play and restrictive-repetitive behaviors. The video-records will be then coded micro-analytically using the Noldus Observer software, to capture moment to moment changes in child behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Irit Mor-Snir, MD, Principal Investigator — Association for Children at Risk
Locations (1):
- Bar Ilan University, Ramat Gan, Israel

REFERENCES:
- [Background] Abidin, R. R. (1995). The Parenting Stress Index Professional Manual. Odessa, FL: Psychological Assessment Resources.
- [Background] Mullen, E. M. (1995). Mullen Scales of Early Learning (AGS ed.). Circle Pines, MN: Circle Pines, MN: American Guidance Service Inc.
- [Background] Rogers, S. J, & Dawson, G. (2010). Early Start Denver Model for Young Children with Autism. Promoting language, learning and engagement. New York: Guilford Press.
- [Background] Johnston, C., & Mash, E. J. (1989). A measure of parenting satisfaction and efficacy. Journal of Clinical Child Psychology, 18(2), 167-175.
- [Background] Sparrow, S. S, Cicchetti, D. V, & Balla, D. A. (2005). Vineland-II Adaptive Behavior Scales: Survey Forms Manual. Circle Pines, MN: AGS Publishing.
- [Background] Davis NO, Carter AS. Parenting stress in mothers and fathers of toddlers with autism spectrum disorders: associations with child characteristics. J Autism Dev Disord. 2008 Aug;38(7):1278-91. doi: 10.1007/s10803-007-0512-z. Epub 2008 Feb 1. PMID 18240012
- [Background] Hall HR, Graff JC. The relationships among adaptive behaviors of children with autism, family support, parenting stress, and coping. Issues Compr Pediatr Nurs. 2011;34(1):4-25. doi: 10.3109/01460862.2011.555270. PMID 21341964
- [Result] Vivanti G, Paynter J, Duncan E, Fothergill H, Dissanayake C, Rogers SJ; Victorian ASELCC Team. Effectiveness and feasibility of the early start denver model implemented in a group-based community childcare setting. J Autism Dev Disord. 2014 Dec;44(12):3140-53. doi: 10.1007/s10803-014-2168-9. PMID 24974255
- [Result] Dawson G, Rogers S, Munson J, Smith M, Winter J, Greenson J, Donaldson A, Varley J. Randomized, controlled trial of an intervention for toddlers with autism: the Early Start Denver Model. Pediatrics. 2010 Jan;125(1):e17-23. doi: 10.1542/peds.2009-0958. Epub 2009 Nov 30. PMID 19948568